CLINICAL TRIAL: NCT04468776
Title: Comparative Effectiveness of Zolpidem/Trazodone and Cognitive Behavioral Therapy for Insomnia in Rural Adults
Brief Title: CBT-I or Zolpidem/Trazodone for Insomnia
Acronym: COZI
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: California Pacific Medical Center Research Institute (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other); University of Pittsburgh (Other); University of Arizona (Other); University of Virginia (Other); University of Illinois at Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CER-2018C2-13262; CER-2018C2-13262 (Other Grant/Funding Number: Patient-Centered Outcomes Research Institute)
Record Dates: First submitted 2020-06-26; First posted 2020-07-13 (Actual); Results first posted 2025-02-24 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Chronic Insomnia
Keywords: Insomnia; Chronic Insomnia; Zolpidem; Ambien; Cognitive-behavioral therapy for insomnia; CBT-I; Rural; Primary Care; Pragmatic Clinical Trial; Comparative Effectiveness; Trazodone
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Zolpidem; Trazodone

STUDY DESIGN:
Intervention Model Description: This study is a randomized (1:1:1) comparative effectiveness trial of medication preference (zolpidem or trazodone), CBT-I, and the combination for the treatment of insomnia in 155 men and women aged 18-80 years living in rural areas.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Masking of participants and providers is not possible given two very different treatment types. The Prime Principal Investigator and a statistician at the Data Coordinating Center will be masked to individual treatment assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Medication (zolpidem or trazodone) (Active Comparator): Zolpidem or trazodone, as prescribed by physician
  Interventions: Drug: Zolpidem; Drug: Trazodone
- Internet Cognitive Behavioral Therapy for Insomnia (CBT-I) (Active Comparator): Internet-based CBT-I program
  Interventions: Behavioral: Internet Cognitive Behavioral Therapy for Insomnia (CBT-I)
- Combination (Experimental): Medication (zolpidem or trazodone) as prescribed by physician and Internet-based CBT-I program
  Interventions: Drug: Zolpidem; Behavioral: Internet Cognitive Behavioral Therapy for Insomnia (CBT-I); Drug: Trazodone

INTERVENTIONS:
Drug: Zolpidem — Zolpidem, as prescribed by physician
  Other Names: Ambien
  Arms: Combination; Medication (zolpidem or trazodone)
Behavioral: Internet Cognitive Behavioral Therapy for Insomnia (CBT-I) — 6-week internet CBT-I multi-component intervention (SHUTi) including sleep restriction, stimulus control, cognitive restructuring, sleep behaviors, and relapse prevention
  Other Names: SHUTi
  Arms: Combination; Internet Cognitive Behavioral Therapy for Insomnia (CBT-I)
Drug: Trazodone — Trazodone, as prescribed by physician
  Other Names: Desyrel
  Arms: Combination; Medication (zolpidem or trazodone)

SUMMARY:
This study is a randomized (1:1:1) comparative effectiveness trial of medication (zolpidem or trazodone), cognitive-behavioral therapy for insomnia (CBT-I), and the combination (medication + CBT-I) for the treatment of chronic insomnia in men and women aged 18-80 living in rural areas with 1 year of follow-up. A total of 155 participants will be enrolled and randomized in the United States. This trial is funded by the Patient-Centered Outcomes Research Institute.

DETAILED DESCRIPTION:
Insomnia is a common health problem that causes distress, impaired function, and increased risk for other health problems. Chronic insomnia is defined by problems with the quality or amount of sleep, including difficulty falling asleep, frequent awakenings, and/or awakening early and being unable to return to sleep. In developing this application, patients, providers, payors, and the investigators identified both concerns and opportunities with current treatments for chronic insomnia. Medications and Cognitive-Behavioral therapy for insomnia (CBT-I; a treatment program to improve sleep through changes in behavior and thinking) are both effective for treating insomnia. Zolpidem, the most frequently prescribed insomnia medication, is widely available, but may cause side effects and dependency. Trazodone is increasingly prescribed off-label for treatment of insomnia, but evidence of efficacy and safety is more limited. CBT-I is the recommended first line treatment by many professional organizations, but it is not widely available in physicians' practices. Patients, providers, and payors face important unanswered questions: Which treatment should be used for the treatment of chronic insomnia? Is combination therapy more effective, and does it result in lower zolpidem use? Who responds best to which treatment? These dilemmas are particularly relevant to patients and providers in rural areas, where access to behavioral health specialists is limited, and concerns regarding use of controlled substances is particularly acute.

To address these questions, we propose the study, Comparative Effectiveness of Zolpidem/Trazodone and Cognitive Behavioral Therapy for Insomnia in Rural Adults (COZI). The investigators will use a well-tested Internet version of CBT-I, which is just as effective as in-person CBT-I, but more widely available. The aims of COZI are to: 1: Compare the effectiveness of medication preference (zolpidem or trazodone), CBT-I, and combination treatment for insomnia symptoms over 6 months. 2: Compare the effectiveness of medication preference, CBT-I, and combination treatment for other symptoms and problems, including health-related quality of life, mood, and health outcomes. 3: Compare the side effects of medication preference, CBT-I, and combination treatment. COZI will study 155 patients recruited from 7 health care systems across the country, each of which has established practices in rural areas. Patients will be treated with medication prescribed by their own physician (zolpidem or trazodone), Internet CBT-I, or a combination of the two. The investigators will evaluate treatment effects at 9 weeks, and 6 and 12 months (with limited additional assessments for adverse events and medication use at 1 and 9 months). Our study questions and design reflect early and ongoing engagement of key stakeholders including patients, providers, and payors, who are members of the Study Advisory Committee (SAC). SAC members will work with study investigators to recommend the best strategies for recruiting patients, measuring treatment effects, and disseminating study findings. The SAC will meet quarterly. Patients and other stakeholders have already provided guidance on which treatments are most worth studying, and which symptoms would best reflect the effects of treatment. Patients and other stakeholders will also be part of the Steering Committee, which is the main decision-making group for our study, and which will meet monthly. COZI will lead to answers for patients and providers addressing insomnia; improved health and function for millions of rural Americans; and sustainable changes in how insomnia is treated in rural practices.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80
* Insomnia Severity Index score > 10
* Regular internet and computer access
* Receives primary care in a Non-metropolitan/Rural residence

Exclusion Criteria:

* Use of hypnotic medication >2 times in the past week
* Current cognitive or cognitive behavioral treatment for insomnia
* Psychotic disorder
* Bipolar disorder
* Current substance use disorder
* Severe Chronic obstructive pulmonary disease (COPD) or other severe pulmonary disease (such as asthma or lung fibrosis)
* Cognitive impairment or dementia
* History of spontaneous or hypnotic-induced complex sleep behavior
* Delayed sleep phase disorder (DSPD)
* Shift work that includes working the night shift (between the hours of 12:00 a.m. - 6:00 a.m.)
* History of fracture or injurious fall in the past 12 months
* Currently pregnant, planning to become pregnant, or breastfeeding
* Other severe or uncontrolled mental or physical disorders that would make participation difficult or unsafe

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 155 (Actual)
Dates: Start 2022-02-25 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Katie L. Stone, PhD, Principal Investigator — California Pacific Medical Center/Sutter Bay Hospitals; Daniel J. Buysse, MD, Principal Investigator — University of Pittsburgh
Locations (7):
- United States (7):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of Arizona, Tucson, Arizona
  - University of Missouri, Columbia, Missouri
  - Oregon Health & Science University, Portland, Oregon
  - Penn State Hershey Medical Center, Hershey, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - University of Virginia, Charlottesville, Virginia

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Medication (Zolpidem or Trazodone) | Internet Cognitive Behavioral Therapy for Insomnia (CBT-I) | Combination
Started | 49 | 54 | 52
9 Weeks Follow-up | 40 | 37 | 41
6 Months Follow-up | 38 | 32 | 34
12 Months Follow-up | 37 | 30 | 33
Completed | 44 | 40 | 43
Not Completed | 5 | 14 | 9
Not completed — Lost to Follow-up | 4 | 3 | 4
Not completed — Withdrawal by Subject | 1 | 10 | 4
Not completed — Physician Decision | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Medication (Zolpidem or Trazodone) | Internet Cognitive Behavioral Therapy for Insomnia (CBT-I) | Combination | Total
Number analyzed (Participants) | 49 | 54 | 52 | 155
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.2 (14.6) | 52.5 (15.3) | 52.5 (15.3) | 53.4 (15.0)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: 1 participant refused to report sex.
  Participants
    number analyzed (Participants) | 49 | 54 | 51 | 154
    Female | 37 | 44 | 37 | 118
    Male | 12 | 10 | 14 | 36
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 3 | 4
  Not Hispanic or Latino | 48 | 54 | 49 | 151
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 3 | 1 | 4
  White | 47 | 49 | 49 | 145
  More than one race | 1 | 1 | 0 | 2
  Unknown or Not Reported | 1 | 0 | 2 | 3
Region of Enrollment [Number; unit: participants]
  United States | 49 | 54 | 52 | 155
Medication preference [Count of Participants; unit: Participants] — Medication preference (zolpidem or trazodone) was determined by the provider and patient. Providers considered factors including patient preference and characteristics (e.g., age, medical and psychiatric history) in their choice of medication. This choice was recorded for each participant before randomization, thereby facilitating unconfounded, randomized comparisons between the three arms. If a participant was randomized to the medication or combination treatment arm, this is the medication that would be prescribed by their provider.
  Participants
    Zolpidem | 11 | 10 | 11 | 32
    Trazodone | 38 | 44 | 41 | 123
Insomnia Severity Index total score [Mean (Standard Deviation); unit: score on a scale] — The Insomnia Severity Index is a 7-item self-report questionnaire that measures severity of insomnia symptoms during the last two weeks. Each item is scored 0 (no problem) to 4 (very severe problem) and the total score ranges 0 to 28, with higher scores indicating more severe insomnia symptoms.
  score on a scale | 18.1 (4.3) | 17.4 (3.7) | 18.9 (4.2) | 18.1 (4.1)

OUTCOME MEASURES:

1. Primary Outcome: Change in Insomnia Symptom Severity
Description: Change in Insomnia Severity Index score from baseline to follow-up. The Insomnia Severity Index is a 7-item self-report questionnaire that measures severity of insomnia symptoms during the last two weeks. Each item is scored 0 (no problem) to 4 (very severe problem) and total between 0-28, with higher scores indicating more severe insomnia symptoms. Change is estimated mean change from mixed-effects linear regression model. Fixed effects: Baseline ISI, Treatment Arm, Visit and Treatment Arm*Visit interaction. Random effects: intercept for Subject, nested within Site.
Time Frame: Baseline, 6 months
Measure: Least Squares Mean (95% Confidence Interval); unit: change score on a scale
Arm/Group | Medication (Zolpidem or Trazodone) | Internet Cognitive Behavioral Therapy for Insomnia (CBT-I) | Combination
Number analyzed (Participants) | 49 | 54 | 52
change score on a scale | -8.05 [-9.44 to -6.65] | -7.82 [-9.32 to -6.32] | -10.19 [-11.66 to -8.73]

2. Secondary Outcome: Number of Participants With Treatment Response of Insomnia Symptoms
Description: Treatment response defined as a ≥6 point reduction in Insomnia Severity Index score from baseline to follow-up. The Insomnia Severity Index is a 7-item self-report questionnaire that measures severity of insomnia symptoms during the last two weeks. Each item is scored 0 (no problem) to 4 (very severe problem) and total between 0-28, with higher scores indicating more severe insomnia symptoms. Data presented as count of participants meeting treatment response criteria at 6 months.
Time Frame: Baseline, 6 months
Population: Only participants who completed the 6 months follow-up assessment were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Medication (Zolpidem or Trazodone) | Internet Cognitive Behavioral Therapy for Insomnia (CBT-I) | Combination
Number analyzed (Participants) | 38 | 32 | 34
Participants | 22 | 21 | 31

3. Secondary Outcome: Number of Participants With Remission of Insomnia Symptoms
Description: Remission of Insomnia symptoms defined as Insomnia Severity Index <8 at follow-up. The Insomnia Severity Index is a 7-item self-report questionnaire that measures severity of insomnia symptoms during the last two weeks. Each item is scored 0 (no problem) to 4 (very severe problem) and total between 0-28, with higher scores indicating more severe insomnia symptoms. Data presented as count of participants meeting insomnia remission criteria at 6 months.
Time Frame: 6 months
Population: Only participants who completed the 6 months follow-up assessment were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Medication (Zolpidem or Trazodone) | Internet Cognitive Behavioral Therapy for Insomnia (CBT-I) | Combination
Number analyzed (Participants) | 38 | 32 | 34
Participants | 16 | 13 | 16

4. Other Pre Specified Outcome: Change in Anxiety and Depression
Description: The Patient Health Questionnaire (PHQ-8) is an 8-item self-report measure for assessing depression severity. The items are summed to yield a score between 0 and 24, with higher scores indicating more frequent depression symptoms.
  The Generalized Anxiety Disorder (GAD-7) Scale is a 7-item self-report measure used for screening and assessing severity of GAD. The items are summed to yield a score between 0 and 21, with higher scores indicating more severe GAD symptoms.
  Change is estimated mean change in mixed-effects linear regression model. Fixed effects: Treatment Arm, Visit and Treatment Arm*Visit interaction. Random effects: intercept for Subject, nested within Site.
Time Frame: Baseline, 6 months
Measure: Least Squares Mean (95% Confidence Interval); unit: change score on a scale
Arm/Group | Medication (Zolpidem or Trazodone) | Internet Cognitive Behavioral Therapy for Insomnia (CBT-I) | Combination
Number analyzed (Participants) | 49 | 54 | 52
change score on a scale
  Patient Health Questionnaire (PHQ-8) | -2.37 [-3.39 to -1.36] | -2.74 [-3.87 to -1.61] | -4.63 [-5.7 to -3.56]
  Generalized Anxiety Disorder (GAD-7) | -1.24 [-2.26 to -0.23] | -2.16 [-3.29 to -1.03] | -2.34 [-3.4 to -1.27]

5. Other Pre Specified Outcome: Change in Cognitive Function
Description: The PROMIS Cognitive Function Short Form (8a) is an 8-item self-report measure related to executive functioning. Individual item responses range from 1 (very often) to 5 (never) and the total raw score is converted to standardized T-scores using established United States general adult population with a mean of 50 and a standard deviation of 10. Higher T-scores signify better cognitive function. Estimated mean change in T-score from baseline to follow-up is reported from mixed-effects linear regression model. Fixed effects: Treatment Arm, Visit and Treatment Arm*Visit interaction. Random effects: intercept for Subject, nested within Site. Positive change indicates improved cognitive function.
Time Frame: Baseline, 6 months
Measure: Least Squares Mean (95% Confidence Interval); unit: T-score
Arm/Group | Medication (Zolpidem or Trazodone) | Internet Cognitive Behavioral Therapy for Insomnia (CBT-I) | Combination
Number analyzed (Participants) | 49 | 54 | 52
T-score | 2.87 [0.81 to 4.93] | 6.64 [4.36 to 8.93] | 4.58 [2.42 to 6.74]

6. Other Pre Specified Outcome: Change in Patient-Reported Health
Description: The PROMIS Global Health is a 10-item self-report measure that assess general health and functioning. Item responses range from 1 (excellent/none) to 5 (poor/always) and a single pain item ranges from 0 (no pain) to 10 (worst pain). Physical and mental health sub-scores are calculated from 4 items each, and the total raw sub-scores (range: 4-20) are converted to T-scores using distributions standardized to mean 50 (SD 10) for the US general population. Higher score indicates greater health-related quality of life.
  The Medical Outcome Survey (SF-12) is a 12-item self-report measure of physical and mental health. The Physical Component Score (PCS) and Mental Component Score (MCS) sub-scores range 0-100; higher score indicates better health.
  Change is estimated mean change from baseline to follow-up in mixed-effects linear regression model. Fixed effects: Treatment Arm, Visit and Treatment Arm*Visit interaction. Random effects: intercept for Subject, nested within Site.
Time Frame: Baseline, 6 months
Measure: Least Squares Mean (95% Confidence Interval); unit: change score on a scale
Arm/Group | Medication (Zolpidem or Trazodone) | Internet Cognitive Behavioral Therapy for Insomnia (CBT-I) | Combination
Number analyzed (Participants) | 49 | 54 | 52
change score on a scale
  Global Health: Mental | 1.22 [-0.52 to 2.95] | 2.43 [0.49 to 4.37] | 4.01 [2.18 to 5.83]
  Global Health: Physical | 2.87 [1.22 to 4.52] | 2.51 [0.68 to 4.35] | 3.59 [1.86 to 5.32]
  SF-12 Physical Component Score | 2.92 [0.75 to 5.09] | 0.07 [-2.33 to 2.46] | 1.92 [-0.34 to 4.18]
  SF-12 Mental Component Score | -0.11 [-2.85 to 2.63] | 4.39 [1.38 to 7.4] | 4.46 [1.61 to 7.3]

7. Other Pre Specified Outcome: Change in Fatigue
Description: The PROMIS Fatigue instrument is a 7-item self-report measure that assesses recent fatigue and how fatigue interfered with daily activities. Scores range from 7 to 35, with higher scores indicating greater fatigue.
  Change is estimated mean change from mixed-effects linear regression model. Fixed effects: Treatment Arm, Visit and Treatment Arm*Visit interaction. Random effects: intercept for Subject, nested within Site.
Time Frame: Baseline, 6 months
Measure: Least Squares Mean (95% Confidence Interval); unit: change score on a scale
Arm/Group | Medication (Zolpidem or Trazodone) | Internet Cognitive Behavioral Therapy for Insomnia (CBT-I) | Combination
Number analyzed (Participants) | 49 | 54 | 52
change score on a scale | -5.44 [-7.99 to -2.89] | -8.82 [-11.66 to -5.99] | -6.8 [-9.48 to -4.12]

8. Other Pre Specified Outcome: Change in Pain Intensity and Interference
Description: The PROMIS Pain Intensity scale is a 3-item instrument used to assess how much pain a person has. Scores range from 3-15, with higher scores indicating greater pain intensity.
  The PROMIS Pain Interference scale is a 6-item instrument used to assess the consequences of pain in different domains of daily life. Scores range from 6-30, with higher scores indicating greater interference.
  Change is estimated mean change from mixed-effects linear regression model. Fixed effects: Treatment Arm, Visit and Treatment Arm*Visit interaction. Random effects: intercept for Subject, nested within Site.
Time Frame: Baseline, 6 months
Measure: Least Squares Mean (95% Confidence Interval); unit: change score on a scale
Arm/Group | Medication (Zolpidem or Trazodone) | Internet Cognitive Behavioral Therapy for Insomnia (CBT-I) | Combination
Number analyzed (Participants) | 49 | 54 | 52
change score on a scale
  Pain Intensity | -0.55 [-2.7 to 1.6] | -1.72 [-4.13 to 0.68] | -3.84 [-6.11 to -1.58]
  Pain Interference | -1.81 [-4.26 to 0.63] | 0.72 [-2.01 to 3.44] | -3.73 [-6.3 to -1.16]

9. Other Pre Specified Outcome: Change in Pittsburgh Sleep Quality Index
Description: The Pittsburgh Sleep Quality Index (PSQI) is an 18-item self-report measure that assesses sleep quality in the past month. These items are combined into seven component scores (subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbance, use of sleep medication, and daytime dysfunction). The seven component scores are added to produce a global sleep quality score ranging from 0 to 21; higher total score indicates worse sleep quality.
  Change is estimated mean change from mixed-effects linear regression model. Fixed effects: Treatment Arm, Visit and Treatment Arm*Visit interaction. Random effects: intercept for Subject, nested within Site.
Time Frame: Baseline, 6 months
Measure: Least Squares Mean (95% Confidence Interval); unit: change score on a scale
Arm/Group | Medication (Zolpidem or Trazodone) | Internet Cognitive Behavioral Therapy for Insomnia (CBT-I) | Combination
Number analyzed (Participants) | 49 | 54 | 52
change score on a scale | -3.42 [-4.46 to -2.38] | -4.52 [-5.67 to -3.37] | -5.23 [-6.32 to -4.15]

10. Other Pre Specified Outcome: Change in Daytime Sleepiness
Description: The Epworth Sleepiness Scale (ESS) is an 8-item self-report measure that assesses daytime sleepiness by asking about the likelihood of dozing in certain situations. Individual items are summed to yield the ESS score between 0 (never doze) to 24 (doze a lot) with higher scores indicating more sleepiness.
  Change is estimated mean change from mixed-effects linear regression model. Fixed effects: Treatment Arm, Visit and Treatment Arm*Visit interaction. Random effects: intercept for Subject, nested within Site.
Time Frame: Baseline, 6 months
Measure: Least Squares Mean (95% Confidence Interval); unit: change score on a scale
Arm/Group | Medication (Zolpidem or Trazodone) | Internet Cognitive Behavioral Therapy for Insomnia (CBT-I) | Combination
Number analyzed (Participants) | 49 | 54 | 52
change score on a scale | -2.81 [-3.77 to -1.84] | -2.61 [-3.68 to -1.54] | -2.18 [-3.2 to -1.17]

11. Other Pre Specified Outcome: Change in Munich Chronotype
Description: The Munich Chronotype Questionnaire (MCTQ) is a self-report scale to assess sleep structure, patterns, duration, and quality. The chronotype sub-score represents the mid-point time of sleep which is converted to a numeric value by adding the hour plus minutes divided by 60. Greater values indicate later chronotype. Positive change values indicate a shift to later chronotype.
  Change is estimated mean change from mixed-effects linear regression model. Fixed effects: Treatment Arm, Visit and Treatment Arm*Visit interaction. Random effects: intercept for Subject, nested within Site.
Time Frame: Baseline, 6 months
Measure: Least Squares Mean (95% Confidence Interval); unit: hours
Arm/Group | Medication (Zolpidem or Trazodone) | Internet Cognitive Behavioral Therapy for Insomnia (CBT-I) | Combination
Number analyzed (Participants) | 49 | 54 | 52
hours | 0.08 [-0.16 to 0.33] | -0.02 [-.029 to 0.24] | 0.23 [-0.03 to 0.5]

12. Other Pre Specified Outcome: Dysfunctional Beliefs and Attitudes About Sleep
Description: Dysfunctional Beliefs and Attitudes about Sleep (DBAS) Scale is a 16-item instrument used to evaluate dysfunctional thoughts related to insomnia. Each item is scored 0-10 and the total is the average of the 16 item scores (range 0-10), with higher scores indicating greater dysfunctional beliefs about sleep.
Time Frame: Baseline, 6 months
Population: 6 months mean only includes those who responded to the DBAS questions on the 6 month follow-up assessment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Medication (Zolpidem or Trazodone) | Internet Cognitive Behavioral Therapy for Insomnia (CBT-I) | Combination
Number analyzed (Participants) | 49 | 54 | 52
score on a scale
  Baseline DBAS mean total score | 6.1 (1.8) | 6.0 (1.3) | 6.2 (1.7)
  6 months DBAS mean total score: number analyzed (Participants) | 38 | 31 | 34
  6 months DBAS mean total score | 5.4 (1.8) | 4.2 (1.6) | 4.0 (2.1)

13. Other Pre Specified Outcome: Number of Participants With Insomnia Treatment Side Effects
Description: Side effects (frequency, severity, impairment) are recorded via self-report adapted from the FIBSER. Scores range from 0 (no side effects; better) to 21 (worse). Side effects were analyzed if participant reported severity of greater than moderate and/or frequency greater than 50% of the time. Count of participants meeting the threshold for analysis up through the 6 month follow-up.
Time Frame: 1 month, 9 weeks, 6 months
Population: Participants included if they completed the 1 month, 9 weeks or 6 month follow-up assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Medication (Zolpidem or Trazodone) | Internet Cognitive Behavioral Therapy for Insomnia (CBT-I) | Combination
Number analyzed (Participants) | 45 | 40 | 41
Participants | 16 | 13 | 15

14. Other Pre Specified Outcome: Medication Adherence
Description: Medication use is assessed using self-reported prescription, over-the-counter, and supplement name and frequency. Count of participants reporting zolpidem or trazodone use for sleep is recorded for adherence to the Medication and Combination treatment arms.
Time Frame: 1 month, 9 weeks, 6 months, 9 months, 12 months
Population: Participants included if they completed the 1 month, 9 weeks, 6 month or 12 month follow-up assessment medications questions.
Measure: Count of Participants; unit: Participants
Arm/Group | Medication (Zolpidem or Trazodone) | Combination
Number analyzed (Participants) | 45 | 44
Participants | 38 | 28

15. Other Pre Specified Outcome: Self-reported Falls
Description: Participants self-reported number of falls including context, location, and consequences of falls. Count of participants with one or more falls up through the 6 month follow-up.
Time Frame: 1 month, 9 weeks, 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Medication (Zolpidem or Trazodone) | Internet Cognitive Behavioral Therapy for Insomnia (CBT-I) | Combination
Number analyzed (Participants) | 49 | 54 | 52
Participants | 8 | 3 | 7

ADVERSE EVENTS:
Time Frame: 12 months
Groups:
- Medication (Zolpidem): Zolpidem: Zolpidem, as prescribed by physician
  Medication preference for zolpidem was recorded prior to randomization by the provider and patient. Patients randomized to the medication arm were prescribed zolpidem by their provider, guided by study-wide recommendations regarding initial doses and dose adjustments, however, prescribers were allowed to use clinical judgment reflecting their usual practice.
- Medication (Trazodone): Trazodone: Trazodone, as prescribed by physician
  Medication preference for trazodone was recorded prior to randomization by the provider and patient. Patients randomized to the medication arm were prescribed trazodone by their provider, guided by study-wide recommendations regarding initial doses and dose adjustments, however, prescribers were allowed to use clinical judgment reflecting their usual practice.
- Combination (Zolpidem): Medication (zolpidem) and Internet-based CBT-I program
  Zolpidem: Zolpidem, as prescribed by physician Medication preference for zolpidem was recorded prior to randomization by the provider and patient. Patients randomized to the medication arm were prescribed zolpidem by their provider, guided by study-wide recommendations regarding initial doses and dose adjustments, however, prescribers were allowed to use clinical judgment reflecting their usual practice.
  Internet Cognitive Behavioral Therapy for Insomnia (CBT-I): 6-week internet CBT-I multi-component intervention (SHUTi) including sleep restriction, stimulus control, cognitive restructuring, sleep behaviors, and relapse prevention
- Combination (Trazodone): Medication (trazodone) and Internet-based CBT-I program
  Trazodone: Trazodone, as prescribed by physician Medication preference for trazodone was recorded prior to randomization by the provider and patient. Patients randomized to the medication arm were prescribed trazodone by their provider, guided by study-wide recommendations regarding initial doses and dose adjustments, however, prescribers were allowed to use clinical judgment reflecting their usual practice.
  Internet Cognitive Behavioral Therapy for Insomnia (CBT-I): 6-week internet CBT-I multi-component intervention (SHUTi) including sleep restriction, stimulus control, cognitive restructuring, sleep behaviors, and relapse prevention
Arm/Group | Medication (Zolpidem) | Medication (Trazodone) | Internet Cognitive Behavioral Therapy for Insomnia (CBT-I) | Combination (Zolpidem) | Combination (Trazodone)
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/38 | 0/54 | 0/11 | 0/41
Serious Adverse Events (participants affected / at risk) | 1/11 | 0/38 | 2/54 | 0/11 | 0/41
Other Adverse Events (participants affected / at risk) | 4/11 | 10/38 | 6/54 | 2/11 | 7/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Medication (Zolpidem) (N=11) | Medication (Trazodone) (N=38) | Internet Cognitive Behavioral Therapy for Insomnia (CBT-I) (N=54) | Combination (Zolpidem) (N=11) | Combination (Trazodone) (N=41)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Medication (Zolpidem) (N=11) | Medication (Trazodone) (N=38) | Internet Cognitive Behavioral Therapy for Insomnia (CBT-I) (N=54) | Combination (Zolpidem) (N=11) | Combination (Trazodone) (N=41)
Palpatations (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 2 | 2 | 0 | 4 — Those who self-reported two or more falls, or a fall resulting in medical care, on scheduled assessments were contacted by the study coordinator to determine causality and outcomes attributed to the event.
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 2 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 1 | 2 | 0 | 0 | 1
Somnolence (Nervous system disorders) | 1 | 6 | 5 | 2 | 3
Confusion (Nervous system disorders) | 1 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-04-20): https://cdn.clinicaltrials.gov/large-docs/76/NCT04468776/Prot_SAP_000.pdf